CLINICAL TRIAL: NCT02018679
Title: Er:YAG Ablative Fractional Laser Assisted-Photodynamic Therapy Versus Photodynamic Therapy for Nodular Basal Cell Carcinoma in Asian: A Prospective, Randomized Study With 12 Months Follow-up
Brief Title: Er:YAG Ablative Fractional Laser Assisted-Photodynamic Therapy Versus Photodynamic Therapy for Basal Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Song Ki-Hoon, Assistant professor and chairman, Department of dermatology Dong-A University, College of medicine, Dong-A University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: DAUDerma-02
Record Dates: First submitted 2013-11-29; First posted 2013-12-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Nodular Basal Cell Carcinoma
Keywords: Nodular basal cell carcinoma; Er:YAG; AFL-assisted; MAL-PDT

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Er:YAG AFL-PDT (Experimental): AFL was performed using a 2940-nm Er:YAG ablative fractional laser (Joule, Sciton Inc., CA, UA) at 550-600 µm ablation in depth, level 1 coagulation, 22% treatment density, and a single pulse. Immediately afterwards, a 1-mm thick layer of MAL (16% Metvix® cream, PhotoCure ASA, Oslo, Norway) was applied to the lesion and to 5 mm of surrounding healthy tissue. The area was covered with an occlusive dressing (Tegaderm, 3M, Saint Paul, MN, US) for 3 hours, after which the remaining cream was removed with saline gauze, and the red fluorescence of porphyrins was visualized with Wood's light. Each treatment area was then separately illuminated with red light-emitting diode (LED) lamps (Aktilite CL128; Galderma, Bruchsal, Germany) with peak emission at 632 nm and total light dose of 37 J cm2.
  Interventions: Procedure: Er:YAG AFL-PDT
- MAL-PDT (Active Comparator): Immediately afterwards, a 1-mm thick layer of MAL (16% Metvix® cream, PhotoCure ASA, Oslo, Norway) was applied to the lesion and to 5 mm of surrounding healthy tissue. The area was covered with an occlusive dressing (Tegaderm, 3M, Saint Paul, MN, US) for 3 hours, after which the remaining cream was removed with saline gauze, and the red fluorescence of porphyrins was visualized with Wood's light. Each treatment area was then separately illuminated with red light-emitting diode (LED) lamps (Aktilite CL128; Galderma, Bruchsal, Germany) with peak emission at 632 nm and total light dose of 37 J cm2. Areas which were scheduled to receive MAL-PDT received the second treatment 7 days later.
  Interventions: Procedure: MAL-PDT

INTERVENTIONS:
Procedure: Er:YAG AFL-PDT — AFL was performed using a 2940-nm Er:YAG ablative fractional laser (Joule, Sciton Inc., CA, UA) at 550-600 µm ablation in depth, level 1 coagulation, 22% treatment density, and a single pulse. Immediately afterwards, a 1-mm thick layer of MAL (16% Metvix® cream, PhotoCure ASA, Oslo, Norway) was applied to the lesion and to 5 mm of surrounding healthy tissue. The area was covered with an occlusive dressing (Tegaderm, 3M, Saint Paul, MN, US) for 3 hours, after which the remaining cream was removed with saline gauze, and the red fluorescence of porphyrins was visualized with Wood's light. Each treatment area was then separately illuminated with red light-emitting diode (LED) lamps (Aktilite CL128; Galderma, Bruchsal, Germany) with peak emission at 632 nm and total light dose of 37 J cm2.
  Arms: Er:YAG AFL-PDT
Procedure: MAL-PDT — a 1-mm thick layer of MAL (16% Metvix® cream, PhotoCure ASA, Oslo, Norway) was applied to the lesion and to 5 mm of surrounding healthy tissue. The area was covered with an occlusive dressing (Tegaderm, 3M, Saint Paul, MN, US) for 3 hours, after which the remaining cream was removed with saline gauze, and the red fluorescence of porphyrins was visualized with Wood's light. Each treatment area was then separately illuminated with red light-emitting diode (LED) lamps (Aktilite CL128; Galderma, Bruchsal, Germany) with peak emission at 632 nm and total light dose of 37 J cm2. Areas which were scheduled to receive MAL-PDT received the second treatment 7 days later.
  Arms: MAL-PDT

SUMMARY:
Topical photodynamic therapy with methyl-aminolaevulinate (MAL-PDT) has been introduced as an alternatively attractive procedure for BCC. Er:YAG ablative fractional laser (AFL) treatment removes the stratum corneum to increase MAL uptake and may improve efficacy. However, no studies have directly compared the efficacy of Er:YAG AFL-PDT and MAL-PDT in treating nodular BCC in Asians.

DETAILED DESCRIPTION:
Basal cell carcinoma (BCC) is the most common cancer in the Caucasian population, with an incidence rising worldwide. there is an increasing trend in the incidence rates of BCC in asian and greater percentage of pigmented BCCs is found to be the most characteristic clinical feature of BCC in Asian compared to BCC in Caucasians. Topical photodynamic therapy with methyl-aminolaevulinate (MAL-PDT) has been introduced as an alternatively attractive procedure for BCC. PDT facilitates the light activation of a photosensitizer in the presence of oxygen. The oxygen generates reactive oxygen species leading to selective and highly localized destruction of abnormal cells. MAL is an efficient photosensitizer as a result of improved lesion penetration attributed to enhanced lipophilicity, decreased charge and also has a greater specificity for neoplastic cells, compared with 5-aminolevulinic acid. Because histologic features of nBCC include down-growth of epithelial buds into the dermis, palisading basal cell and separation of epidermis from the underlying dermis, it is generally treated twice within an interval of 1 week.But, MAL-PDT shows the lower efficacy for the treatment of pigmented BCC because melanin disturbs the absorption of the MAL. Also, a significantly higher proportions of BCC in the Asian population were pigmented BCC compared with pigmented BCC of Caucasian. Consequently, additional techniques are needed to enhance the penetration and accumulation of MAL in order to improve PDT efficacy and decrease treatment duration in darker-skinned patients.

Er:YAG ablative fractional laser therapy (AFL) can ablate the epidermis and dermis without significant thermal injury. This approach creates microscopic ablation zones (MAZ) in laser-applied portion of the skin. The tissue with MAZ is surrounded by thin layers of coagulated tissue. Since the Er:YAG AFL resurfaces 5-20% of the skin at one time and does not injure the entire thickness of the epidermis, healing times are minimized. Recent studies have demonstrated that Er:YAG AFL facilitates delivery and uptake of topical MAL deep into the skin, enhancing porphyrin synthesis and photodynamic activation. We have compared the efficacy, recurrence rate, cosmetic outcomes and safety of Er:YAG AFL-PDT with standard MAL-PDT in the treatment of nBCC among Korean populations.

ELIGIBILITY:
Inclusion Criteria:

* patient's request for alternative treatment due to the lower cosmetic outcomes of surgery
* difficulty to surgical excision due to bleeding abnormalities or cardiac problems

Exclusion Criteria:

* patients with more than 5 eligible lesions
* lesions deeper than 2mm in depth
* lesions located in the midface region, nose, orbital areas, and ears
* lesions with a longest diameter of less than 6 mm or more than 15mm
* infiltrative BCC
* morpheaform BCC
* known allergies to the MAL cream or lidocaine
* pregnancy
* lactation
* any active systemic infectious disease
* immunosuppressive treatment
* personal history of malignant melanoma
* tendency towards melasma or keloid formation
* prior treatment of the lesions within 4 weeks
* any indication of poor compliance

Ages: 38 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-03; Primary Completion 2013-02 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Difference the efficacy between Er:YAG AFL-PDT and MAL-PDT | Efficacy was evaluated at 3 months and 12 months after treatment
  Lesion responses were classified as either a complete response (complete disappearance of the lesion) or a non-complete response (incomplete disappearance)

SECONDARY OUTCOMES:
Difference of the cosmetic outcomes between Er:YAG AFL-PDT and MAL-PDT treatment | Cosmetic outcome was assessed by each investigator for all lesions that achieved a complete response at 3 or 12 months
  I was graded using a 4-point scale: excellent (only slight occurrence of redness or change in pigmentation), good (moderate redness or change in pigmentation), fair (slight to moderate scarring, atrophy, or induration), or poor (extensive scarring, atrophy, or induration)

OTHER OUTCOMES:
Difference of the recurrence rates between Er:YAG AFL-PDT and MAL-PDT | recurrence rates were evaluated at 12 months after the last treatment.
  In all cases of complete response, the patients were reviewed at 12 months to check for recurrence. Recurrence was assessed by inspection, dermoscopy, photography, palpation, and histologic findings.
Difference of the safety between Er:YAG AFL-PDT and MAL-PDT | Safety assessments were performed at the end of the 3-hour cream application; after the illumination during each treatment session; and at 1 week, 3 months, and 12 months after the last treatment
  Adverse events reported by the patient were noted at each follow-up visit, including severity, duration, and need for additional treatment.
  The severity of the adverse event was assessed as follows: mild (transient and easily tolerated); moderate (caused the patient discomfort and interrupted usual activities); and severe (caused considerable interference with usual activities and may have been incapacitating or life threatening).
  All adverse events due to PDT were described as phototoxic reactions (i.e. erythema, postinflammatory hyperpigmentation, edema, itching, oozing, bleeding, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Hoon Song, M.D., Ph.D., Study Chair — Dong-A University
Locations (1):
- Dong-A University, Busan, Seo-gu, South Korea